CLINICAL TRIAL: NCT05291819
Title: A NORwegian Randomized Strategy Trial in PsoRiatic Arthritis: ImagiNg Treat-to-target vs Conventional Treat-to-target
Brief Title: Imaging Treat-to-target Strategy vs Conventional Treat-to-target Strategy in Psoriatic Arthritis
Acronym: NOR-SPRINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Siri Lillegraven, Principal Investigator, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOR-SPRINT protocol ver4_1
Record Dates: First submitted 2022-03-02; First posted 2022-03-23 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Psoriatic Arthritis
Keywords: Imaging; Treat-to-target
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Intervention Model Description: A two-arm, parallel-group, single-blind, treatment strategy study where patients are randomized 1:1 to a conventional treat-to-target follow-up strategy with structured clinical assessment of disease activity or an imaging informed treat-to-target follow-up strategy with both structured clinical assessment of disease activity and structured imaging assessment of disease activity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treat-to-target (Other): Conventional treat-to-target follow-up strategy with structured clinical assessment of disease activity
  Interventions: Other: Conventional treat-to-target
- Imaging informed treat-to-target (Experimental): Imaging informed treat-to-target follow-up strategy with both structured clinical assessment of disease activity and structured imaging assessment of disease activity.
  Interventions: Other: Imaging informed treat-to-target

INTERVENTIONS:
Other: Imaging informed treat-to-target — A treat-to-target treatment strategy incorporating information from ultrasound assessment of joints, tendons and entheses (at every visit), and magnetic resonance imaging (MRI) of spine and sacroiliac (SI)-joints at baseline and 1 year, in addition to clinical information
  Specifically, this means that these additional measures will be added to conventional treat to target:
  * If evidence of enthesitis (power Doppler>0 in enthesis) or axial inflammation (SPARCC score ≥ 2* in SI-joint or SPARCC score ≥ 5 in presence of clinical symptoms of axial disease) on imaging the patient will progress directly to biological disease modifying antirheumatic drug in the treatment algorithm
  * If evidence of ongoing inflammation (power Doppler>0) on ultrasound assessment of joints, tendons or enthesis, the patient will be classified as not having reached their treatment target
  Arms: Imaging informed treat-to-target
Other: Conventional treat-to-target — Patients are treated according to an algorithm based on current European recommendations. The conventional treatment target, applicable to both arms and the target in the conventional arm, is all of: Disease Activity index in PSoriatic Arthritis (DAPSA) remission (≤4), Enthesitis ≤1, Psoriasis Body Surface Area ≤3%
  Arms: Conventional treat-to-target

SUMMARY:
The main objective is to assess if a treat-to-target strategy implementing structured imaging assessments leads to better patient outcome in terms of sustained remission compared to a conventional treat-to-target strategy in psoriatic arthritis.

Main inclusion criteria are: >18 years of age, Clinical diagnosis of psoriatic arthritis (PsA), Fulfillment of ClASsification of Psoriatic Arthritis (CASPAR) criteria, Indication for treatment with disease modifying anti-rheumatic drugs according to treating physician

Primary endpoint: Sustained remission, defined as Very Low Disease Activity (VLDA) at 16, 20 and 24 months

Secondary endpoints: Individual and composite disease activity measures and remission criteria, inflammation assessed by ultrasound, health related quality of life and adverse events.

Study design: A two-arm, parallel-group, single-blind, treatment strategy study where patients are randomized 1:1 to a conventional treat-to-target follow-up strategy with structured clinical assessment of disease activity or an imaging informed treat-to-target follow-up strategy with both structured clinical assessment of disease activity and structured imaging assessment of disease activity. Duration of follow-up is 24 months.

All patients are treated according to an algorithm based on current European recommendations. The conventional treatment target, applicable to both arms and the sole target in the conventional arm, is all of: Disease Activity index in Psoriatic Arthritis (DAPSA) remission (≤3), Enthesitis ≤1, Psoriasis Body Surface Area ≤3%

Intervention: A treat-to-target treatment strategy incorporating information from ultrasound assessment of joints, tendons and entheses (at every visit), and magnetic resonance imaging (MRI) of spine and sacroiliac (SI)-joints at baseline and 1 year, in addition to clinical information. Specifically, this means that these additional measures will be added to conventional treat to target:

* If evidence of enthesitis or axial inflammation on imaging the patient will progress directly to biological disease modifying antirheumatic drug in the treatment algorithm
* If evidence of ongoing inflammation (power Doppler>0) on ultrasound assessment of joints, tendons or enthesis, the patient will be classified as not having reached their treatment target

DETAILED DESCRIPTION:
This project addresses the challenges associated with psoriatic arthritis (PsA), which is a diverse disease which is difficult to assess clinically. Ultrasound and magnetic resonance imaging (MRI) visualize inflammation that is not apparent on clinical examination, but whether treating patients according to these findings improves outcomes is unknown.

The main objective is to assess if a treat-to-target strategy implementing structured imaging assessments leads to better patient outcome in terms of sustained remission compared to a conventional treat-to-target strategy in psoriatic arthritis.

Primary endpoint: Sustained remission, defined as Very Low Disease Activity (VLDA) at all of the 16, 20 and 24 month visits.

Secondary endpoints include Individual and composite disease activity measures and remission criteria, inflammation assessed by ultrasound, health related quality of life and adverse events.

Study design: A two-arm, parallel-group, single-blind, treatment strategy study where patients are randomized 1:1 to a conventional treat-to-target follow-up strategy with structured clinical assessment of disease activity or an imaging informed treat-to-target follow-up strategy with both structured clinical assessment of disease activity and structured imaging assessment of disease activity. Duration of follow-up is 24 months.

All patients are treated according to an algorithm based on current European recommendations. The conventional treatment target, applicable to both arms and the sole target in the conventional arm, is all of: Disease Activity index in Psoriatic Arthritis (DAPSA) remission (≤3), Enthesitis ≤1, Psoriasis Body Surface Area ≤3%

Intervention: A treat-to-target treatment strategy incorporating information from ultrasound assessment of joints, tendons and entheses (at every visit), and magnetic resonance imaging (MRI) of spine and sacroiliac (SI)-joints at baseline and 1 year, in addition to clinical information. Specifically, this means that these additional measures will be added to conventional treat to target:

If evidence of enthesitis or axial inflammation on imaging the patient will progress directly to biological disease modifying antirheumatic drug in the treatment algorithm If evidence of ongoing inflammation (power Doppler>0) on ultrasound assessment of joints, tendons or enthesis, the patient will be classified as not having reached their treatment target

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>18 years of age)
2. Clinical diagnosis of PsA
3. Indication for treatment with DMARDs according to treating physician (including having attempted ≥2 non-steroidal anti-inflammatory drugs (NSAIDs) for a minimum of 4 weeks in total in predominantly axial and/or entheseal disease)
4. Fulfillment of CASPAR criteria for PsA

Exclusion Criteria:

1. Verified arthritis >1 year prior to inclusion
2. Previous DMARD treatment for PsA
3. Systemic glucocorticoid use within the last 3 months
4. Local glucocorticoid injections within the last 4 weeks
5. Major co-morbidities, including but not limited to relevant malignancies, severe diabetes mellitus, severe infections, uncontrolled hypertension, severe cardiovascular disease (NYHA class III or IV) and/or severe respiratory diseases and cirrhosis.
6. Indications of active or latent tuberculosis (TB) as assessed by chest radiograph and TB interferon gamma release assay (IGRA). Patients with documented adequately treated latent TB can be included.
7. Any other medical condition that according to the treated physician and/or local guidelines makes adherence to treatment protocol impossible
8. Abnormal renal function, defined as serum creatinine >142 µmol/L in female and >168 µmol/L in male, or estimated glomerular filtration rate (eGFR) <40 mL/min/1.73 m2
9. Abnormal liver function (defined as Aspartate Transaminase (AST) and/or Alanine Transaminase (ALT) >1.5 x upper normal limit), active or recent hepatitis
10. Significant anemia, leukopenia and/or thrombocytopenia
11. Inadequate birth control, pregnancy, and/or breastfeeding (current at screening or planned within the duration of the study)
12. Contraindications to magnetic resonance imaging
13. Severe psychiatric or mental disorders, alcohol abuse or other substance abuse, language barriers or other factors which makes adherence to the study protocol impossible
14. Established or suspected widespread-pain syndrome/fibromyalgia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sustained Remission | Sustained remission is defined by the patient meeting VLDA at all of 16, 20 and 24 month follow-up visits
  Sustained remission defined as a combination of Very Low Disease Activity (VLDA) at all of the time points 16, 20 and 24 months.
  VLDA requires all of the following to be met: Tender joint count (68) ≤ 1, swollen joint count (66) ≤ 1, Psoriasis Body Surface Area ≤ 3, Enthesitis≤ 1, Patient global assessment of disease severity VAS (0-100) ≤ 20, Pain VAS (0-100) ≤ 15 and Health Assessment Questionnaire Disability Index ≤ 0.5.

SECONDARY OUTCOMES:
Patient global assessment of disease activity | 12 and 24 months
  Patient global assessment of disease activity on a 0-100 visual analogue scale (VAS), with higher scores Indicating more disease activity
Patient pain assessment | 12 and 24 months
  Patient pain assessment on a 0-100 visual analogue scale, with higher scores Indicating more pain
Patient fatigue assessment | 12 and 24 months
  Patient fatigue assessment on a 0-100 visual analogue scale, with higher scores Indicating more fatigue
66 joint count for swollen joints | 12 and 24 months
  Structured 66 joint count for swollen joints
68 joint count for tender joints | 12 and 24 months
  Structured 68 joint count for tender joints
Tender dactylitis count | 12 and 24 months
  Structured tender dactylitis count
Spondyloarthritis Research Consortium of Canada Enthesitis Index (SPARCC entheseal index) | 12 and 24 months
  SPARCC magnetic resonance imaging entheseal index
Body surface area of skin psoriasis | 12 and 24 months
  Body surface area of skin psoriasis in percentage
Modified Nail Psoriasis Severity Index (mNAPSI) | 12 and 24 months
  Modified Nail Psoriasis Severity Index (mNAPSI)
Physician global assessment of disease activity | 12 and 24 months
  Physician global assessment of disease activity on a 0-100 visual analogue scale, with higher scores Indicating more disease activity
C-reactive protein (CRP) | 12 and 24 months
  C-reactive protein (CRP), higher scores indicating more inflammation
Erythrocyte sedimentation rate (ESR) | 12 and 24 months
  Erythrocyte sedimentation rate (ESR), higher scores indicating more inflammation
Disease activity in Psoriatic arthritis Score (DAPSA) | 12 and 24 months
  Disease activity in Psoriatic arthritis Score (DAPSA), higher scores indicating more disease activity
Minimal Disease Activity (MDA) | 12 and 24 months
  Minimal Disease Activity (MDA). MDA is a composite assessment of disease activity state in PsA. It includes 7 components: tender joint count (68) ≤ 1, swollen joint count (66) ≤ 1, Psoriasis Area Severity Index ≤ 1/Body Surface Area ≤ 3, enthesitis≤ 1, patient global assessment of disease activity VAS ≤ 20, pain VAS ≤ 15 and HAQ-DI ≤ 0.5. MDA requires 5 out of 7 components to be met.
Psoriatic Arthritis Disease Activity Score (PASDAS) | 12 and 24 months
  Psoriatic Arthritis Disease Activity Score (PASDAS) is a composite disease activity index, with higher scores indicating more disease activity
American College of Rheumatology (ACR) 20 response | 12 and 24 months
  American College of Rheumatology (ACR) 20 response is defined as ≥ 20 % improvement in swollen and tender joint counts plus ≥ 20 % improvement in 3 of the 5 remaining ACR core set variables; pain VAS, physician global VAS, Health Assessment Questionnaire Disability Index (HAQ-DI) and CRP/ESR.
Structured assessment of joints by musculoskeletal ultrasound according to a predefined protocol | 12 and 24 months
  Structured assessment of joints by musculoskeletal ultrasound according to a predefined protocol
Structured assessment of entheses by musculoskeletal ultrasound according to a predefined protocol | 12 and 24 months
  Structured assessment of entheses by musculoskeletal ultrasound according to a predefined protocol
Structured assessment of tendons by musculoskeletal ultrasound according to a predefined protocol | 12 and 24 months
  Structured assessment of tendons by musculoskeletal ultrasound according to a predefined protocol
Health Related Quality of Life | 12 and 24 months
  Assessed by Short Form 36 (SF-36) questionnaire
Adverse events | 0-24 months
  Number and nature of adverse events and serious adverse events

OTHER OUTCOMES:
Patient global assessment of disease activity | 0-24 months
  Patient global assessment of disease activity on a 0-100 visual analogue scale, with higher scores Indicating more disease activity
Patient pain assessment | 0-24 months
  Patient pain assessment on a 0-100 visual analogue scale, with higher scores Indicating more pain
Patient fatigue assessment | 0-24 months
  Patient fatigue assessment on a 0-100 visual analogue scale, with higher scores Indicating more fatigue
Bath Ankylosing Spondylitis Disease Activity Index | 0-24 months
  Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), higher scores indicating more disease activity
Patient acceptable symptom state | 0-24 months
  Patient acceptable symptom state (PASS)
66 joint count for swollen joints | 0-24 months
  66 joint count for swollen joints
68 joint count for tender joints | 0-24 months
  68 joint count for tender joints
Tender dactylitis count | 0-24 months
  Tender dactylitis count
Spondyloarthritis Research Consortium of Canada Enthesitis Index (SPARCC entheseal index) | 0-24 months
  SPARCC MRI entheseal index
Body surface area of skin psoriasis | 0-24 months
  Body surface area of skin psoriasis in percentages
Investigator global assessment of skin psoriasis | 0-24 months
  Investigator global assessment of skin psoriasis
Modified Nail Psoriasis Severity Index (mNAPSI) | 0-24 months
  Modified Nail Psoriasis Severity Index (mNAPSI)
Physician global assessment of disease activity | 0-24 months
  Physician global assessment of disease activity on a 0-100 visual analogue scale
C-reactive protein (CRP) | 0-24 months
  C-reactive protein (CRP), higher scores indicating more inflammation
Erythrocyte sedimentation rate (ESR) | 0-24 months
  Erythrocyte sedimentation rate (ESR), higher scores indicating more inflammation
Disease activity in Psoriatic arthritis Score (DAPSA) | 0-24 months
  Disease activity in Psoriatic arthritis Score (DAPSA)
Minimal Disease Activity (MDA) | 0-24 months
  Minimal Disease Activity (MDA). MDA is a composite assessment of disease activity state in PsA. It includes 7 components: tender joint count (68) ≤ 1, swollen joint count (66) ≤ 1, Psoriasis Area Severity Index ≤ 1/Body Surface Area ≤ 3, enthesitis≤ 1, patient global assessment of disease activity VAS ≤ 20, pain VAS ≤ 15 and HAQ-DI ≤ 0.5. MDA requires 5 out of 7 components to be met.
Psoriatic Arthritis Disease Activity Score (PASDAS) | 0-24 months
  Psoriatic Arthritis Disease Activity Score (PASDAS) is a composite disease activity index, with higher scores indicating more disease activity
American College of Rheumatology (ACR) response | 0-24 months
  American College of Rheumatology (ACR) response
Disease Activity score 28 (DAS-28) | 0-24 months
  Disease Activity score 28 (DAS-28)
Inflammation assessed musculoskeletal ultrasound | 0 and 24 months
  1. Joints (as specified in protocol)
  2. Entheses (as specified in protocol)
  3. Tendons (as specified in protocol)
  4. Peritenonitis (as specified in protocol)
Inflammation assessed by MRI | 12 and 24 months
  MRI of total spine and sacroiliac joint, assessed by SPARCC score
Joint damage assessed by radiography of hands and feet | 24 months
  Assessed by the modified Sharp van der Heijde Score
Work Productivity and Activity Impairment Questionnaire (WPAI) | 0-24 months
  Work Productivity and Activity Impairment Questionnaire (WPAI)
Work participation | 0-24 months
  Work participation based on data from Statistics Norways's event database (FD Trygd) (social benefits)
Euro Quality of Life 5 Dimensions (EQ-5D) | 0-24 months
  Euro Quality of Life 5 Dimensions (EQ-5D)
Short Form 36 (SF-36) | 0-24 months
  Short Form 36 (SF-36)
Psoriatic Arthritis Impact of Disease (PsAID) | 0-24 months
  Psoriatic Arthritis Impact of Disease (PsAID)
Health Assessment Questionnaire Disability Index (HAQ-DI) | 0-24 months
  Health Assessment Questionnaire Disability Index (HAQ-DI)
Use of hospital services | 0-24 months
  Use of hospital services from The Norwegian Patient Register
Medication prescription | 0-24 months
  Prescription of medication from The Norwegian Prescription Register (pharmaceuticals)
Use of primary care resources | 0-24 months
  Use of primary care resources based on data from Norway Control and Payment of Health Reimbursement (KUHR) database (primary care services) (d) Municipal patient- and user register (IPLOS) database (nursing services)
Use of nursing services | 0-24 months
  Use of nursing services based on the municipal patient- and user register (IPLOS) database

CONTACTS AND LOCATIONS:
Overall Officials: Siri Lillegraven, MD, MPH, PhD, Principal Investigator — Diakonhjemmet
Locations (12):
- Norway (12):
  - Department of Rheumatology, Helse Møre og Romsdal HF, Ålesund
  - Department of Rheumatology, Haukeland University Hospital, Helse Bergen HF, Bergen
  - Department of Rheumatology, Drammen Hospital, Vestre Viken HF, Drammen
  - Helse Førde, Førde
  - Haugesunds Sanitetsforening Revmatismesykehus, Haugesund
  - Sørlandet Sykehus, Kristiansand
  - Revmatismesykehuset AS, Lillehammer
  - Helgelandssykehuset, Mo i Rana, Mo i Rana
  - Department of Rheumatology, Diakonhjemmet Hospital, Oslo
  - Martina Hansens Hospital AS, Sandvika
  - University Hospital of Northern Norway, Tromsø
  - Department of Rheumatology, St Olavs Hospital HF, Trondheim